CLINICAL TRIAL: NCT01493297
Title: Effects of Vitamin A and Carotenoids on Iron Absorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Instituto Venezolano de Investigaciones Cientificas (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Principal investigator, Swiss Federal Institute of Technology
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: ETH-FeVZ
Record Dates: First submitted 2011-11-29; First posted 2011-12-15 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Iron Absorption
Keywords: Retinyl palmitate, beta-carotene, stable isotopes, radio isotopes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Retinyl palmitate (Other): Labeled iron as FeSO4 (4 mg) added to a test meal with or without retinyl palmitate (1000 RE)
  Interventions: Other: Labeled iron solutions
- Beta-carotene (Other): Labeled iron as FeSO4 (4 mg) added to a test meal with or without beta-carotene (1000 RE)
  Interventions: Other: Labeled iron solutions

INTERVENTIONS:
Other: Labeled iron solutions — Labeled iron as FeSO4 (4 mg/test meal)

SUMMARY:
The objective of this study is to investigate the effect of vitamin A and carotenoids on iron absorption in healthy subjects with low and normal vitamin A status. Vitamin A and carotenoids have been reported to enhance the nonheme iron absorption, but the results from human isotope studies are equivocal. Radio-iron studies in Venezuelan adults have consistently reported an increase in iron absorption, whereas stable and radio isotopes studies conducted in Sweden and Switzerland reported no influence. Differences in vitamin A status of the subjects may be a possible explanation for the contradictory findings. In this study, iron absorption will be measured from an iron-fortified maize bread meal with or without retinyl palmitate or β-carotene by using both stable- and radioactive-isotope techniques in Venezuelan women with a range of vitamin A status.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-52 years old
* Body weight ≤ 70 kg
* Body mass index (BMI), 18.5-30 kg/m2
* Adequate vitamin A status (SR ≥ 0.7 μmol/L, n=20)
* Inadequate vitamin A status (SR < 0.7 μmol/L, n=20)
* No major medical illnesses (no known infection, gastrointestinal or metabolic disorders)

Exclusion Criteria:

* Pregnancy or lactation
* Regular intake of medication (except oral contraceptives)
* Blood donation or significant blood loss (accident, surgery) over the past 4 months
* Currently participating in another clinical trial or having participated in another clinical trial during the last 3 months prior to the beginning of this study
* Former participation in a study involving administration of iron stable isotopes

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Fractional iron absorption | 1 month after enrollment
  Iron absorption will be estimated by measuring the erythrocyte incorporation of stable (57Fe/58Fe) and radio (55Fe/59Fe) iron isotopes labels given in test meals.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Andersson, Dr, Principal Investigator — Swiss Federal Institute of Technology, ETH Zurich
Locations (1):
- Venezuelan Institute for Scientific Research (IVIC), Caracas, Venezuela

REFERENCES:
- [Background] Walczyk T, Davidsson L, Rossander-Hulthen L, Hallberg L, Hurrell RF. No enhancing effect of vitamin A on iron absorption in humans. Am J Clin Nutr. 2003 Jan;77(1):144-9. doi: 10.1093/ajcn/77.1.144. PMID 12499334
- [Background] Garcia-Casal MN, Layrisse M, Solano L, Baron MA, Arguello F, Llovera D, Ramirez J, Leets I, Tropper E. Vitamin A and beta-carotene can improve nonheme iron absorption from rice, wheat and corn by humans. J Nutr. 1998 Mar;128(3):646-50. doi: 10.1093/jn/128.3.646. PMID 9482776
- [Background] Garcia-Casal MN. Carotenoids increase iron absorption from cereal based food in the human. Nutr Res 2006;26:340-4.
- [Background] Layrisse M, Garcia-Casal MN, Solano L, et al. The role of vitamin A on the inhibitors of nonheme iron absorption: preliminary results. J Nutr Biochem 1997;8:61-7.